CLINICAL TRIAL: NCT04908189
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Deucravacitinib in Participants With Active Psoriatic Arthritis (PsA) Who Are Naïve to Biologic Disease Modifying Anti-rheumatic Drugs or Had Previously Received TNFα Inhibitor Treatment
Brief Title: A Study to Determine the Efficacy and Safety of Deucravacitinib Compared With Placebo in Participants With Active Psoriatic Arthritis (PsA) Who Are Naïve to Biologic Disease Modifying Anti-rheumatic Drugs or Had Previously Received TNFα Inhibitor Treatment
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-055; 2020-005099-36 (EudraCT Number); U1111-1259-9466 (Registry Identifier: WHO)
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis; PsA; Deucravacitinib; BMS-986165; Apremilast; Otezla
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — deucravacitinib; apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Deucravacitinib (Experimental)
  Interventions: Drug: Deucravacitinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Deucravacitinib; Other: Placebo
- Apremilast (Other)
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: BMS-986165
  Arms: Deucravacitinib; Placebo
Other: Placebo — Specified dose on specified days
  Arms: Placebo
Drug: Apremilast — Specified dose on specified days
  Other Names: Otezla
  Arms: Apremilast

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of deucravacitinib versus placebo for the treatment of participants with active PsA who are naïve to biologic disease modifying antirheumatic drugs or had previously received TNFα inhibitor treatment.The long term extension period will provide additional long-term safety and efficacy information.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed to have psoriatic arthritis (PsA) of at least 3 months duration at Screening
* Meets the Classification Criteria for Psoriatic Arthritis (CASPAR) criteria at Screening
* Active plaque psoriatic skin lesion(s) or documented medical history of plaque psoriasis (PsO) at Screening
* Active arthritis as shown by ≥ 3 swollen joints and ≥ 3 tender joints at Screening and Day 1
* Participant has high sensitivity C-reactive protein (hsCRP) ≥ 3 mg/L at Screening
* Must have completed the week 52 treatment for the optional open-label long-term extension period

Exclusion Criteria:

* Nonplaque psoriasis at Screening or Day 1
* Other autoimmune condition such as systemic lupus erythematous, mixed connective tissue disease, multiple sclerosis, or vasculitis
* History of or current inflammatory joint disease other than PsA (e.g., gout, reactive arthritis, rheumatoid arthritis, ankylosing spondylitis, Lyme disease)
* Active fibromyalgia
* Received an approved or investigational biologic therapy for the treatment of PsA or PsO

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 729 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2026-11-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (138):
- United States (24):
  - Local Institution - 0149, Mountain Brook, Alabama
  - Local Institution - 0212, Sacramento, California
  - Local Institution - 0188, Whittier, California
  - Local Institution - 0192, Skokie, Illinois
  - Local Institution - 0203, Hopkinsville, Kentucky
  - Local Institution - 0195, Baton Rouge, Louisiana
  - Local Institution - 0169, Cumberland, Maryland
  - Local Institution - 0034, Okemos, Michigan
  - Local Institution - 0133, Eagan, Minnesota
  - Local Institution - 0109, Hattiesburg, Mississippi
  - Local Institution - 0108, New York, New York
  - Local Institution - 0186, Rochester, New York
  - Local Institution - 0196, Charlotte, North Carolina
  - Local Institution - 0180, Cleveland, Ohio
  - Local Institution - 0189, Oklahoma City, Oklahoma
  - Local Institution - 0147, Portland, Oregon
  - Local Institution - 0016, Duncansville, Pennsylvania
  - Local Institution - 0182, Summerville, South Carolina
  - Local Institution - 0167, Lubbock, Texas
  - Local Institution - 0070, Mesquite, Texas
  - Local Institution - 0184, Plano, Texas
  - Local Institution - 0187, Seattle, Washington
  - Local Institution - 0190, Franklin, Wisconsin
  - Local Institution - 0175, Milwaukee, Wisconsin
- Argentina (5):
  - Local Institution - 0048, La Plata, Buenos Aires
  - Local Institution - 0038, San Isidro, Buenos Aires
  - Local Institution - 0039, CABA, Distrito Federal
  - Local Institution - 0171, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0200, Buenos Aires
- Australia (6):
  - Local Institution - 0003, Botany, New South Wales
  - Local Institution - 0018, Paramatta, New South Wales
  - Local Institution - 0004, Maroochydore, Queensland
  - Local Institution - 0099, Woodville, South Australia
  - Local Institution - 0002, Camberwell, Victoria
  - Local Institution - 0017, Geelong, Victoria
- Belgium (3):
  - Local Institution - 0078, Brussels
  - Local Institution - 0058, Ghent
  - Local Institution - 0061, Liège
- Canada (5):
  - Local Institution - 0111, Vancouver, British Columbia
  - Local Institution - 0006, Hamilton, Ontario
  - Local Institution - 0030, Markham, Ontario
  - Local Institution - 0036, Toronto, Ontario
  - Local Institution - 0001, Québec
- China (25):
  - Local Institution - 0126, Bengbu, Anhui
  - Local Institution - 0152, Beijing, Beijing Municipality
  - Local Institution - 0146, Beijing, Beijing Municipality
  - Local Institution - 0153, Guangzhou, Guangdong
  - Local Institution - 0135, Guangzhou, Guangdong
  - Local Institution - 0206, Shenzhen, Guangdong
  - Local Institution - 0127, Zhengzhou, Henan
  - Local Institution - 0170, Changsha, Hunan
  - Local Institution - 0161, Changsha, Hunan
  - Local Institution - 0125, Changzhou, Jiangsu
  - Local Institution - 0138, Nanjing, Jiangsu
  - Local Institution - 0139, Nantong, Jiangsu
  - Local Institution - 0163, Wuxi, Jiangsu
  - Local Institution - 0148, Jiujiang, Jiangxi
  - Local Institution - 0131, Nanchang, Jiangxi
  - Local Institution - 0156, Nanchang, Jiangxi
  - Local Institution - 0140, Pingxiang, Jiangxi
  - Local Institution - 0158, Baotou, Neimeng
  - Local Institution - 0157, Hohhot, Neimeng
  - Local Institution - 0154, Xi'an, Shan3xi
  - Local Institution - 0207, Shanghai, Shanghai Municipality
  - Local Institution - 0164, Chengdu, Sichuan
  - Local Institution - 0117, Ürümqi, Xinjiang
  - Local Institution - 0134, Kunming, Yunnan
  - Local Institution - 0129, Wenzhou, Zhejiang
- Colombia (5):
  - Local Institution - 0072, Barranquilla, Atlántico
  - Local Institution - 0015, Bogotá
  - Local Institution - 0020, Cali
  - Local Institution - 0022, Chía
  - Local Institution - 0019, Medellín
- Czechia (5):
  - Local Institution - 0010, Brno
  - Local Institution - 0009, Ostrava
  - Local Institution - 0035, Ostrava
  - Local Institution - 0011, Prague
  - Local Institution - 0023, Uherské Hradiště
- Germany (7):
  - Local Institution - 0176, Ratingen, North Rhine-Westphalia
  - Local Institution - 0101, Cologne
  - Local Institution - 0199, Erlangen
  - Local Institution - 0046, Hamburg
  - Local Institution - 0075, Magdeburg
  - Local Institution - 0201, Minden
  - Local Institution - 0074, Tübingen
- Hungary (6):
  - Local Institution - 0025, Veszprém, Veszprém City
  - Local Institution - 0197, Budapest
  - Local Institution - 0066, Debrecen
  - Local Institution - 0028, Gyula
  - Local Institution - 0024, Hódmezővásárhely
  - Local Institution - 0027, Kistarcsa
- Italy (3):
  - Azienda Ospedaliera Universitaria Careggi-Reumatologia, Florence
  - AOR San Carlo di Potenza-UOC Reumatologia, Potenza
  - Local Institution - 0097, Roma
- Japan (15):
  - Local Institution - 0202, Nagoya, Aichi-ken
  - Local Institution - 0106, Nagoya, Aichi-ken
  - Local Institution - 0151, Sapporo, Hokkaido
  - Local Institution - 0179, Tsu, Mie-ken
  - Local Institution - 0123, Kawachi-Nagano, Osaka
  - Local Institution - 0205, Bunkyō, Tokyo
  - Local Institution - 0121, Chuo-ku, Tokyo
  - Local Institution - 0067, Itabashi-ku, Tokyo
  - Local Institution - 0178, Meguro-ku, Tokyo
  - Local Institution - 0122, Minato-ku, Tokyo
  - Local Institution - 0174, Mitaka, Tokyo
  - Local Institution - 0065, Shinjuku-ku, Tokyo
  - Local Institution - 0155, Fukuoka
  - Local Institution - 0166, Osaka
  - Local Institution - 0204, Osaka
- Mexico (6):
  - Local Institution - 0052, León, Guanajuato
  - Local Institution - 0051, Guadalajara, Jalisco
  - Local Institution - 0057, Zapopan, Jalisco
  - Local Institution - 0198, Mexico City, Mexico City
  - Local Institution - 0056, Mérida, Yucatán
  - Local Institution - 0053, Chihuahua City
- Poland (6):
  - Local Institution - 0082, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0177, Warsaw, Masovian Voivodeship
  - Local Institution - 0079, Gdansk, Pomeranian Voivodeship
  - Local Institution - 0080, Elblag
  - Local Institution - 0081, Torun
  - Local Institution - 0112, Wroclaw
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Novosibirsk
- Spain (4):
  - Local Institution - 0014, Barcelona
  - Local Institution - 0012, Madrid
  - Local Institution - 0045, Santander
  - Local Institution - 0013, Valencia
- Taiwan (5):
  - Local Institution - 0090, Taichung
  - Local Institution - 0088, Taichung
  - Local Institution - 0089, Taichung
  - Local Institution - 0091, Taipei
  - Local Institution - 0087, Taipei
- United Kingdom (6):
  - Local Institution - 0185, London, England
  - Local Institution - 0060, Bradford
  - Local Institution - 0064, Hull
  - Local Institution - 0077, Liverpool
  - Local Institution - 0062, London
  - Local Institution - 0105, Manchester

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04908189.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Deucravacitinib: Deucravacitinib 6 mg daily
- Placebo: Placebo daily
- Apremilast: Apremilast 30 mg twice daily
Period: Pre-treatment
Arm/Group | Deucravacitinib | Placebo | Apremilast
Started (Randomized) | 312 | 312 | 105
Completed (Treated) | 312 | 311 | 105
Not Completed | 0 | 1 | 0
Period: Placebo-Controlled (Week 0 - Week 16)
Arm/Group | Deucravacitinib | Placebo | Apremilast
Started | 312 | 311 | 105
Completed | 292 | 292 | 90
Not Completed | 20 | 19 | 15
Not completed — Lack of Efficacy | 1 | 3 | 0
Not completed — Adverse Event | 6 | 4 | 10
Not completed — Participant request to discontinue study treatment | 2 | 4 | 2
Not completed — Withdrawal by Subject | 6 | 8 | 3
Not completed — Administrative reason by sponsor | 3 | 0 | 0
Not completed — Other reasons | 2 | 0 | 0
Period: Active Treatment (Week 16 - Week 52)
Arm/Group | Deucravacitinib | Placebo | Apremilast
Started | 292 | 292 | 90
Participants Switched to Deucravacitinib | 0 | 292 | 0
Completed | 266 | 269 | 79
Not Completed | 26 | 23 | 11
Not completed — Lack of Efficacy | 6 | 6 | 1
Not completed — Adverse Event | 9 | 7 | 3
Not completed — Participant request to discontinue study treatment | 3 | 3 | 4
Not completed — Withdrawal by Subject | 5 | 5 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Other reasons | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deucravacitinib | Placebo | Apremilast | Total
Number analyzed (Participants) | 312 | 312 | 105 | 729
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.7 (11.73) | 49.3 (12.18) | 49.1 (13.47) | 49.0 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 168 | 56 | 377
  Male | 159 | 144 | 49 | 352
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 50 | 16 | 120
  Not Hispanic or Latino | 195 | 200 | 64 | 459
  Unknown or Not Reported | 63 | 62 | 25 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 7 | 4 | 24
  Asian | 54 | 45 | 28 | 127
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 223 | 240 | 65 | 528
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 22 | 19 | 8 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting American College of Rheumatology (ACR) 20 at Week 16
Description: The American College of Rheumatology (ACR) 20 is defined as 20% improvement over baseline in tender (68) and swollen (66) joint counts and a 20% improvement in 3 of the 5 remaining core data set measures: Participant Global Assessment of Disease Activity; Participant Global Assessment of Pain; Participant assessment of physical function; Physician Global Assessment of psoriatic arthritis; and Acute phase reactant value of high sensitivity C-reactive protein (hsCRP). Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 312 | 312
Participants | 169 | 123

2. Secondary Outcome: Change From Baseline in Disease Activity Score 28 C-reactive Protein (DAS28-CRP) at Week 16
Description: DAS28-CRP is a composite of how many joints in the hands (including metacarpophalangeal and proximal interphalangeal joints but excluding DIPs), wrists, elbows, shoulders, and knees are swollen and/or tender out of a total of 28; CRP in the blood to measure the degree of inflammation, and participant global assessment of disease activity. The results are combined to produce the DAS28-CRP score that range from 1.0 to 9.4, which correlates with the extent of disease activity: < 2.6=disease remission; 2.6 - 3.2=low disease activity; 3.2-5.1=moderate disease activity; >5.1=high disease activity. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in DAS28-CRP indicates an improvement.
Time Frame: Baseline, Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with DAS28-CRP baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 300 | 299
score on a scale | -1.3133 (1.17420) | -0.9095 (1.10470)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted Mean Difference = -0.4743, 95% CI 2-sided [-0.6455 to -0.3031], Standard Error of Mean 0.08735 — The adjusted mean difference and p-value are based on the total randomized population, which is 312 for Deucravacitinib and 312 for Placebo

3. Secondary Outcome: Change From Baseline in Health Assessment Quiestionnaire - Disability Index (HAQ-DI) at Week 16
Description: HAQ-DI is a patient-reported outcome measure that assesses the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2 to 3 items. For each item in the questionnaire, the level of activity is scored from 0 to 3, with 0 representing "no difficulty," 1 representing "some difficulty," 2 representing "much difficulty," and 3 representing "unable to do." increasing scores for the 8 disability categories indicate increasing level of difficulty. HAQDI is calculated by summing the adjusted categories scores and dividing by the number of categories answered. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in HAQ-DI indicates an improvement.
Time Frame: Baseline, Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with HAQ-DI baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 307 | 311
score on a scale | -0.3103 (0.46159) | -0.2219 (0.46858)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Test type: Superiority; p = 0.0013, ANCOVA; Adjusted mean difference = -0.1126, 95% CI 2-sided [-0.1814 to -0.0438], Standard Error of Mean 0.03511 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Participants Meeting Psoriasis Area and Severity Index 75 (PASI 75) at Week 16
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 is the number of participants who experience at least a 75% improvement in PASI score as compared with the baseline value. Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: Week 16
Population: All randomized participants of deucravacitinib and placebo with at least 3% body surface area (BSA) and at least static physician's global assessment (sPGA) 2 at baseline as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 154 | 149
Participants | 63 | 23

5. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Physical Component Summary (PCS) Score at Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The physical component summary (PCS) consists of these 4 subscales: Physical functioning, Role-physical, Bodily pain, General health. The scores range from 0 to 100, with a higher score indicating better quality of life. The PCS summary scores will be calculated by taking a weighted linear combination of the individual subscales. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 PCS indicates an improvement.
Time Frame: Baseline, Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with SF-36 PCS baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 307 | 310
Score on a scale | 6.194 (7.4640) | 4.262 (7.0328)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Test type: Superiority; p = 0.0002, ANCOVA; Adjusted mean difference = 2.042, 95% CI 2-sided [0.980 to 3.105], Standard Error of Mean 0.5421 — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Number of Participants Meeting Enthesitis Resolution (Score of 0) Among Participants With Enthesitis at Baseline by Leeds Enthesitis Index (LEI) at Week 16
Description: Number of participants meeting enthesitis resolution (score of 0) among participants with enthesitis at Baseline by Leeds Enthesitis Index (LEI). An overall score of 0 to 6 is derived from the presence or absence of tenderness at 6 enthesial sites (right and left: lateral epicondyle, medial femoral condyle, and Achilles tendon insertion) at the time of evaluation. A higher count indicates a greater enthesitis burden.
Time Frame: Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with enthesitis at baseline by LEI
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 140 | 150
Participants | 74 | 66

7. Secondary Outcome: Number of Participants Meeting Achievement of Minimal Disease Activity (MDA) at Week 16
Description: Number participants meeting achievement of MDA where an MDA response is achievement of 5 of 7 following outcomes at Week 16:
  1. Tender joint count ≤ 1
  2. Swollen joint count ≤ 1
  3. Psoriasis Area and Severity Index (PASI) ≤ 1 or body surface area (BSA) ≤ 3%
  4. Patient assessment of psoriatic arthiritis (PsA) pain ≤ 15
  5. Patient Global Assessment of PsA disease activity ≤ 20
  6. HAQ-DI ≤ 0.5
  7. Tender enthesial points ≤ 1
Time Frame: Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 312 | 312
Participants | 80 | 46

8. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score at Week 16
Description: FACIT-Fatigue evaluates a range of self-reported symptoms over the past week, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience or symptoms of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. The recall period is 7 days. Each item is rated on a 5-point Likert scale ranging from 0 = "not at all" to 4 = "very much." Sum scores for the 13 items range from 0 through 52, where higher scores indicate less fatigue. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in FACIT-Fatigue indicates an improvement.
Time Frame: Baseline, Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with FACIT-Fatigue baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 307 | 310
Score on a scale | 2.6 (8.17) | 1.9 (8.54)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Test type: Superiority; p = 0.2017, ANCOVA; Adjusted mean difference = 0.8, 95% CI 2-sided [-0.4 to 2.0], Standard Error of Mean 0.61 — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Number of Participants Meeting Dactylitis Resolution at Week 16
Description: Number of participants meeting dactylitis resolution at Week 16 among the participants with dactylitis at baseline, where resolution is defined as a tender dactylitis count of 0 in participants with a tender dactylitis count ≥ 1 at baseline. The number of digits in hands and feet with dactylitis will be counted by a blinded assessor.
Time Frame: Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with tender dactylitis count >=1 at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 78 | 80
Participants | 43 | 36

10. Secondary Outcome: Number of Participants Meeting American College of Rheumatology (ACR) 50 at Week 16
Description: The American College of Rheumatology (ACR) 50 is defined as 50% improvement over baseline in tender (68) and swollen (66) joint counts and a 50% improvement in 3 of the 5 remaining core data set measures: Participant Global Assessment of Disease Activity; Participant Global Assessment of Pain; Participant assessment of physical function; Physician Global Assessment of psoriatic arthritis; and Acute phase reactant value of high sensitivity C-reactive protein (hsCRP). Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 312 | 312
Participants | 90 | 51

11. Secondary Outcome: Number of Participants Meeting American College of Rheumatology (ACR) 70 at Week 16
Description: The American College of Rheumatology (ACR) 70 is defined as 70% improvement over baseline in tender (68) and swollen (66) joint counts and a 70% improvement in 3 of the 5 remaining core data set measures: Participant Global Assessment of Disease Activity; Participant Global Assessment of Pain; Participant assessment of physical function; Physician Global Assessment of psoriatic arthritis; and Acute phase reactant value of high sensitivity C-reactive protein (hsCRP). Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 312 | 312
Participants | 33 | 17

12. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: as for outcome 3
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 309 | 311
score on a scale
  Week 2: number analyzed (Participants) | 307 | 309
  Week 2 | -0.0546 (0.38637) | -0.1335 (0.34583)
  Week 4: number analyzed (Participants) | 307 | 309
  Week 4 | -0.1547 (0.41308) | -0.1760 (0.40042)
  Week 8: number analyzed (Participants) | 308 | 310
  Week 8 | -0.2301 (0.44365) | -0.1964 (0.43603)
  Week 12: number analyzed (Participants) | 309 | 308
  Week 12 | -0.2544 (0.45565) | -0.2236 (0.46098)
  Week 16: number analyzed (Participants) | 307 | 311
  Week 16 | -0.3103 (0.46159) | -0.2219 (0.46858)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 2; Test type: Superiority; p = 0.0231, ANCOVA; Adjusted mean difference = 0.0643, 95% CI 2-sided [0.0088 to 0.1198], Standard Error of Mean 0.02831 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 4; Test type: Superiority; p = 0.7865, ANCOVA; Adjusted mean difference = 0.0085, 95% CI 2-sided [-0.0528 to 0.0697], Standard Error of Mean 0.03126 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 8; Test type: Superiority; p = 0.1280, ANCOVA; Adjusted mean difference = -0.0515, 95% CI 2-sided [-0.1179 to 0.0148], Standard Error of Mean 0.03386 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Deucravacitinib vs Placebo; Week 12; Test type: Superiority; p = 0.1180, ANCOVA; Adjusted mean differnce = -0.0541, 95% CI 2-sided [-0.1219 to 0.0137], Standard Error of Mean 0.03460 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Deucravacitinib vs Placebo; Week 16; Test type: Superiority; p = 0.0013, ANCOVA; Adjusted mean difference = -0.1126, 95% CI 2-sided [-0.1814 to -0.0438], Standard Error of Mean 0.03511 — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Number of Participants Who Achieve a Clinically Meaningful Improvement in HAQ-DI Score at Week 16
Description: Number of participants who achieve a clinically meaningful improvement (≥ 0.35 improvement from baseline) in HAQ-DI score among participants with a HAQ-DI score ≥ 0.35 at baseline. HAQ-DI is a patient-reported outcome measure that assesses the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2 to 3 items. For each item in the questionnaire, the level of activity is scored from 0 to 3, with 0 representing "no difficulty," 1 representing "some difficulty," 2 representing "much difficulty," and 3 representing "unable to do." increasing scores for the 8 disability categories indicate increasing level of difficulty. HAQDI is calculated by summing the adjusted categories scores and dividing by the number of categories answered.
Time Frame: Week 16
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 268 | 273
Participants | 131 | 118

14. Secondary Outcome: Number of Participants Meeting Psoriasis Area and Severity Index 75 (PASI 75)
Description: as for outcome 4
Time Frame: Weeks 4, 8, 12, 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 154 | 149
Participants
  Week 4 | 14 | 10
  Week 8 | 26 | 19
  Week 12 | 45 | 22
  Week 16 | 63 | 23

15. Secondary Outcome: Number of Participants Meeting Psoriasis Area and Severity Index 90 (PASI 90)
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 90 is the number of participants who experience at least a 90% improvement in PASI score as compared with the baseline value. Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: Weeks 4, 8, 12, 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 154 | 149
Participants
  Week 4 | 4 | 3
  Week 8 | 10 | 7
  Week 12 | 31 | 15
  Week 16 | 41 | 13

16. Secondary Outcome: Number of Participants Meeting Psoriasis Area and Severity Index 100 (PASI 100)
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 100 is the number of participants who experience at least a 100% improvement in PASI score as compared with the baseline value. Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: Weeks 4, 8, 12, 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 154 | 149
Participants
  Week 4 | 2 | 0
  Week 8 | 6 | 3
  Week 12 | 17 | 9
  Week 16 | 24 | 8

17. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Physical Component Summary (PCS) Score
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 12, 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 308 | 310
Score on a scale
  Week 4: number analyzed (Participants) | 307 | 308
  Week 4 | 3.364 (5.8439) | 2.771 (5.8897)
  Week 12: number analyzed (Participants) | 308 | 307
  Week 12 | 5.419 (7.1066) | 3.578 (6.7537)
  Week 16: number analyzed (Participants) | 307 | 310
  Week 16 | 6.194 (7.4640) | 4.262 (7.0328)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 4; Test type: Superiority; p = 0.1147, ANCOVA; Adjusted mean difference = 0.692, 95% CI 2-sided [-0.168 to 1.551], Standard Error of Mean 0.4384 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 12; Test type: Superiority; p = 0.0001, ANCOVA; Adjusted mean difference = 1.999, 95% CI 2-sided [0.991 to 3.008], Standard Error of Mean 0.5147 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 16; Test type: Superiority; p = 0.0002, ANCOVA; Adjusted mean difference = 2.042, 95% CI 2-sided [0.980 to 3.105], Standard Error of Mean 0.5421 — [estimate comment as in outcome 2, analysis 1]

18. Secondary Outcome: Number of Participants Meeting Enthesitis Resolution (Score of 0) Among Participants With Enthesitis at Baseline by Leeds Enthesitis Index (LEI)
Description: as for outcome 6
Time Frame: Weeks 4, 8, 12, 16
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 140 | 150
Participants
  Week 4: number analyzed (Participants) | 137 | 148
  Week 4 | 45 | 55
  Week 8: number analyzed (Participants) | 138 | 147
  Week 8 | 70 | 54
  Week 12: number analyzed (Participants) | 138 | 147
  Week 12 | 74 | 58
  Week 16 | 74 | 66

19. Secondary Outcome: Number of Participants Meeting Enthesitis Resolution (Score of 0) Among Participants With Enthesitis at Baseline by Spondyloarthritis Research Consortium of Canada (SPARCC)
Description: Number of participants meeting enthesitis resolution (score of 0) among participants with enthesitis at Baseline by SPARCC. The SPARCC Enthesitis Index has a 0 to 16 score that is derived from the evaluation of 8 locations: the greater trochanter (right [R]/left [L]), quadriceps tendon insertion into the patella (R/L), patellar ligament insertion into the patella and tibial tuberosity (R/L), Achilles tendon insertion (R/L), plantar fascia insertion (R/L), medial and lateral epicondyles (R/L), and supraspinatus insertion (R/L). A higher count indicates a higher enthesitis burden based on the current evaluation.
Time Frame: Weeks 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with enthesitis at baseline by SPARCC
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 177 | 196
Participants
  Week 4 | 53 | 55
  Week 8 | 73 | 55
  Week 12 | 75 | 66
  Week 16 | 86 | 75

20. Secondary Outcome: Number of Participants Meeting Achievement of Minimal Disease Activity (MDA)
Description: as for outcome 7
Time Frame: Weeks 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 312 | 312
Participants
  Week 4 | 19 | 16
  Week 8 | 35 | 28
  Week 12 | 56 | 24
  Week 16 | 80 | 46

21. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Mental Component Summary (MCS) Score
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The mental component summary (MCS) of the SF-36 consists of these 4 subscales: Vitality, Social functioning, Role-emotional, Mental health. The scores range from 0 to 100, with a higher score indicating better quality of life. The MCS summary scores will be calculated by taking a weighted linear combination of the individual subscales. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 MCS indicates an improvement.
Time Frame: Baseline, Weeks 4, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with SF-36 MCS baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 308 | 310
Score on a scale
  Week 4: number analyzed (Participants) | 307 | 308
  Week 4 | 0.195 (7.7026) | 0.300 (7.7067)
  Week 12: number analyzed (Participants) | 308 | 307
  Week 12 | 1.245 (8.6442) | 0.123 (9.1804)
  Week 16: number analyzed (Participants) | 307 | 310
  Week 16 | 1.009 (9.7740) | -0.438 (9.3388)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 4; Test type: Superiority; p = 0.6159, ANCOVA; Adjusted mean difference = -0.284, 95% CI 2-sided [-1.396 to 0.827], Standard Error of Mean 0.5670 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 12; Test type: Superiority; p = 0.1847, ANCOVA; Adjusted mean difference = 0.829, 95% CI 2-sided [-0.396 to 2.054], Standard Error of Mean 0.6250 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 16; Test type: Superiority; p = 0.0888, ANCOVA; Adjusted mean difference = 1.145, 95% CI 2-sided [-0.174 to 2.464], Standard Error of Mean 0.6730 — [estimate comment as in outcome 2, analysis 1]

22. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score
Description: as for outcome 8
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 309 | 310
Score on a scale
  Week 2: number analyzed (Participants) | 307 | 308
  Week 2 | 0.8 (6.60) | 1.5 (6.52)
  Week 4: number analyzed (Participants) | 307 | 308
  Week 4 | 1.3 (6.70) | 1.6 (6.95)
  Week 8: number analyzed (Participants) | 308 | 309
  Week 8 | 2.9 (7.53) | 1.9 (8.54)
  Week 12: number analyzed (Participants) | 309 | 307
  Week 12 | 2.2 (8.40) | 2.0 (8.91)
  Week 16: number analyzed (Participants) | 307 | 310
  Week 16 | 2.6 (8.17) | 1.9 (8.54)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 2; Test type: Superiority; p = 0.1924, ANCOVA; Adjusted mean difference = -0.6, 95% CI 2-sided [-1.6 to 0.3], Standard Error of Mean 0.49 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 4; Test type: Superiority; p = 0.7601, ANCOVA; Adjusted mean difference = -0.2, 95% CI 2-sided [-1.20 to 0.8], Standard Error of Mean 0.51 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 8; Test type: Superiority; p = 0.0303, ANCOVA; Adjusted mean difference = 1.3, 95% CI 2-sided [0.1 to 2.4], Standard Error of Mean 0.59 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Deucravacitinib vs Placebo; Week 12; Test type: Superiority; p = 0.4747, ANCOVA; Adjusted mean difference = 0.5, 95% CI 2-sided [-0.8 to 1.7], Standard Error of Mean 0.63 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Deucravacitinib vs Placebo; Week 16; Test type: Superiority; p = 0.2017, ANCOVA; Adjusted mean difference = 0.8, 95% CI 2-sided [-0.4 to 2.0], Standard Error of Mean 0.61 — [estimate comment as in outcome 2, analysis 1]

23. Secondary Outcome: Number of Participants Meeting Dactylitis Resolution
Description: as for outcome 9
Time Frame: Weeks 4, 8, 12, 16
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 78 | 80
Participants
  Week 4 | 24 | 30
  Week 8 | 31 | 27
  Week 12 | 39 | 29
  Week 16 | 43 | 36

24. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Impact of Disease (PsAID) 12 Score
Description: The Psoriatic Arthritis Impact of Disease (PsAID) is a 12-item self-report that measures PsA symptoms and impact of disease. Each item is scored on a 0 to 10 numeric rating scale with a 1-week recall period. The PsAID has a total score, with a higher value indicating worse health. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in PsAID indicates an improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 309 | 310
Score on a scale
  Week 2: number analyzed (Participants) | 307 | 308
  Week 2 | -0.658 (1.3895) | -0.590 (1.2369)
  Week 4: number analyzed (Participants) | 307 | 308
  Week 4 | -0.986 (1.5902) | -0.761 (1.5206)
  Week 8: number analyzed (Participants) | 308 | 309
  Week 8 | -1.419 (1.7445) | -0.849 (1.8018)
  Week 12: number analyzed (Participants) | 309 | 307
  Week 12 | -1.511 (1.9314) | -0.937 (1.9126)
  Week 16: number analyzed (Participants) | 307 | 310
  Week 16 | -1.729 (2.0150) | -0.968 (1.9075)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 2; Test type: Superiority; p = 0.4459, ANCOVA; Adjusted mean difference = -0.077, 95% CI 2-sided [-0.276 to 0.122], Standard Error of Mean 0.1015 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 4; Test type: Superiority; p = 0.0461, ANCOVA; Adjusted mean difference = -0.232, 95% CI 2-sided [-0.460 to -0.004], Standard Error of Mean 0.1164 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 8; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -0.598, 95% CI 2-sided [-0.857 to -0.339], Standard Error of Mean 0.1321 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Deucravacitinib vs Placebo; Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -0.605, 95% CI 2-sided [-0.882 to -0.327], Standard Error of Mean 0.1416 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Deucravacitinib vs Placebo; Week 16; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -0.786, 95% CI 2-sided [-1.071 to -0.501], Standard Error of Mean 0.1455 — [estimate comment as in outcome 2, analysis 1]

25. Secondary Outcome: Change From Baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) Score
Description: The Disease Activity Index for Psoriatic Arthritis Score is a composite measure to assess peripheral joint involvement that is based upon numerical summation of 5 variables of disease activity: tender joint count (0-68), swollen joint count (0-66), Participant Global Assessment of Disease Activity (0 to 10 cm VAS, 0= excellent and 10= poor), Participant Global Assessment of Pain (0 to 10 centimeter [cm] visual analog scale (VAS), 0= no pain, 10= worst possible pain), and C-reactive protein. A higher DAPSA score indicated more active disease activity. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in DAPSA indicates an improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with DAPSA baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 308 | 307
Score on a scale
  Week 2: number analyzed (Participants) | 307 | 306
  Week 2 | -4.9619 (12.27319) | -5.9569 (12.24097)
  Week 4: number analyzed (Participants) | 302 | 304
  Week 4 | -9.0129 (11.93271) | -8.2813 (12.79788)
  Week 8: number analyzed (Participants) | 303 | 301
  Week 8 | -13.5855 (14.33402) | -10.7292 (16.10715)
  Week 12 | -15.7385 (16.02197) | -11.8980 (16.33187)
  Week 16: number analyzed (Participants) | 300 | 299
  Week 16 | -17.5225 (16.66002) | -12.1547 (17.74566)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 2; Test type: Superiority; p = 0.7025, ANCOVA; Adjusted mean difference = 0.3525, 95% CI 2-sided [-1.4560 to 2.1609], Standard Error of Mean 0.92270 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 4; Test type: Superiority; p = 0.1413, ANCOVA; Adjusted mean difference = -1.3730, 95% CI 2-sided [-3.2023 to 0.4562], Standard Error of Mean 0.93331 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 8; Test type: Superiority; p = 0.0007, ANCOVA; Adjused mean difference = -3.7522, 95% CI 2-sided [-5.9155 to -1.5890], Standard Error of Mean 1.10374 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Deucravacitinib vs Placebo; Week 12; Test type: Superiority; p < 0.0001, ANOVA; Adjusted mean difference = -4.8072, 95% CI 2-sided [-7.0388 to -2.5757], Standard Error of Mean 1.13857 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Deucravacitinib vs Placebo; Week 16; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -6.2006, 95% CI 2-sided [-8.6082 to -3.7930], Standard Error of Mean 1.22840 — [estimate comment as in outcome 2, analysis 1]

26. Secondary Outcome: Number of Participants With Achievement of Disease Activity Index for Psoriatic Arthritis (DAPSA) Low Disease Activity Response
Description: The Disease Activity Index for Psoriatic Arthritis Score is a composite measure to assess peripheral joint involvement that is based upon numerical summation of 5 variables of disease activity: tender joint count (0-68), swollen joint count (0-66), Participant Global Assessment of Disease Activity (0 to 10 cm VAS, 0= excellent and 10= poor), Participant Global Assessment of Pain (0 to 10 centimeter [cm] visual analog scale (VAS), 0= no pain, 10= worst possible pain), and C-reactive protein. A higher DAPSA score indicated more active disease activity.
Time Frame: Weeks 2, 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 312 | 312
Participants
  Week 2 | 25 | 18
  Week 4 | 44 | 42
  Week 8 | 69 | 55
  Week 12 | 95 | 66
  Week 16 | 104 | 78

27. Secondary Outcome: Number of Participants With Achievement of Disease Activity Index for Psoriatic Arthritis (DAPSA) Disease Remission
Description: as for outcome 26
Time Frame: Weeks 2, 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 312 | 312
Participants
  Week 2 | 1 | 1
  Week 4 | 2 | 1
  Week 8 | 12 | 4
  Week 12 | 20 | 8
  Week 16 | 30 | 9

28. Secondary Outcome: Number of Participants Meeting Achievement of Physician Global Assessment-Fingernails (PGA-F) of 0/1
Description: The overall condition of the fingernails is rated on a 5-point scale: 0 = clear, 1 = minimal, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: Weeks 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with a baseline PGA-F score of >= 3
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 51 | 45
Participants
  Week 4 | 10 | 10
  Week 8 | 13 | 13
  Week 12 | 16 | 11
  Week 16 | 17 | 15

29. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) 28 C-reactive Protein (CRP) Score
Description: The DAS28-CRP is a composite outcome measure that assesses: 1) How many joints in the hands (including metacarpophalangeal and proximal interphalangeal joints but excluding DIPs), wrists, elbows, shoulders, and knees are swollen and/or tender out of a total of 28; 2) CRP in the blood to measure the degree of inflammation; 3) Participant Global Assessment of Disease Activity. DAS28-CRP scores range from 1.0 to 9.4, where lower scores indicate less disease activity. The results are combined to produce the DAS28-CRP score, which correlates with the extent of disease activity: < 2.6: Disease remission, 2.6 to 3.2: Low disease activity, 3.2 to 5.1: Moderate disease activity, > 5.1: High disease activity. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in DAS28-CRP indicates an improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 308 | 307
Score on a scale
  Week 2: number analyzed (Participants) | 307 | 306
  Week 2 | -0.3226 (0.74392) | -0.4044 (0.70334)
  Week 4: number analyzed (Participants) | 302 | 304
  Week 4 | -0.6292 (0.84069) | -0.5888 (0.75652)
  Week 8: number analyzed (Participants) | 303 | 301
  Week 8 | -0.9992 (1.01750) | -0.7579 (0.99991)
  Week 12 | -1.1279 (1.14379) | -0.8826 (1.03604)
  Week 16: number analyzed (Participants) | 300 | 299
  Week 16 | -1.3133 (1.17420) | -0.9095 (1.10470)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 2; Test type: Superiority; p = 0.5707, ANCOVA; Adjusted mean difference = 0.0318, 95% CI 2-sided [-0.0782 to 0.1419], Standard Error of Mean 0.05613 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 4; Test type: Superiority; p = 0.1862, ANCOVA; Adjusted mean difference = -0.0833, 95% CI 2-sided [-0.2069 to 0.0402], Standard Error of Mean 0.06303 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 8; Test type: Superiority; p = 0.0002, ANCOVA; Adjusted mean difference = -0.2958, 95% CI 2-sided [-0.4497 to -0.1418], Standard Error of Mean 0.07854 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Deucravacitinib vs Placebo; Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -0.3262, 95% CI 2-sided [-0.4889 to -0.1635], Standard Error of Mean 0.08300 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Deucravacitinib vs Placebo; Week 16; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -0.4743, 95% CI 2-sided [-0.6455 to -0.3031], Standard Error of Mean 0.08735 — [estimate comment as in outcome 2, analysis 1]

30. Secondary Outcome: Number of Participants With Achievement of Disease Activity Score (DAS) 28 C-reactive Protein (CRP) Low Disease Activity Response
Description: The DAS28-CRP is a composite outcome measure that assesses: 1) How many joints in the hands (including metacarpophalangeal and proximal interphalangeal joints but excluding DIPs), wrists, elbows, shoulders, and knees are swollen and/or tender out of a total of 28; 2) CRP in the blood to measure the degree of inflammation; 3) Participant Global Assessment of Disease Activity. DAS28-CRP scores range from 1.0 to 9.4, where lower scores indicate less disease activity. The results are combined to produce the DAS28-CRP score, which correlates with the extent of disease activity: < 2.6: Disease remission, 2.6 to 3.2: Low disease activity, 3.2 to 5.1: Moderate disease activity, > 5.1: High disease activity.
Time Frame: Weeks 2, 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 312 | 312
Participants
  Week 2 | 23 | 19
  Week 4 | 39 | 31
  Week 8 | 35 | 32
  Week 12 | 54 | 39
  Week 16 | 56 | 43

31. Secondary Outcome: Number of Participants With Achievement of Disease Activity Score (DAS) 28 C-reactive Protein (CRP) Disease Remission
Description: as for outcome 30
Time Frame: Weeks 2, 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 312 | 312
Participants
  Week 2 | 13 | 7
  Week 4 | 27 | 14
  Week 8 | 57 | 31
  Week 12 | 64 | 35
  Week 16 | 84 | 44

32. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Disease Activity Score (PASDAS)
Description: The Psoriatic Arthritis Disease Activity Score (PASDAS) is a composite measure calculated from the Physician Global Assessment of PsA, the Participant Global Assessment of Disease Activity, the Short Form-36 PCS, the swollen joint count, the tender joint count, the Enthesitis (LEI), the Dactylitis (LDI) (Basic), and the High-sensitivity C-reactive protein (hsCRP). The range of PASDAS is 0-10. Higher score means more active disease. Change from baseline is defined as value at post-baseline visit. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Weeks 4, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with PASDAS baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 306 | 305
Score on a scale
  Week 4: number analyzed (Participants) | 299 | 300
  Week 4 | -0.8037 (0.90993) | -0.7690 (0.90884)
  Week 12 | -1.5273 (1.27441) | -1.0137 (1.17400)
  Week 16: number analyzed (Participants) | 300 | 297
  Week 16 | -1.7047 (1.32902) | -1.1434 (1.26434)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 4; Test type: Superiority; p = 0.2836, ANCOVA; Adjusted mean difference = -0.0758, 95% CI 2-sided [-0.2144 to 0.0627], Standard Error of Mean 0.07069 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -0.5548, 95% CI 2-sided [-0.7396 to -0.3699], Standard Error of Mean 0.09431 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 16; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -0.5835, 95% CI 2-sided [-0.7826 to -0.3843], Standard Error of Mean 0.10162 — [estimate comment as in outcome 2, analysis 1]

33. Secondary Outcome: Change From Baseline in Modified Composite Psoriatic Disease Activity Index (mCPDAI)
Description: Four domains are used to calculate the modified Composite Psoriatic Disease Activity Index (mCPDAI): joints (66 swollen joint count and 68 tender joint count; Health Assessment Questionnaire), skin (PASI and DLQI), dactylitis (a simple count of each digit involved), and enthesitis (number of tendons/fascia insertion sites showing enthesitis scored from 0 to 4, based on palpation of Achilles tendon and bilateral plantar fasciae insertion). The mCPDAI is scored using a 4 point scale from 0 (no disease activity) to 3 (most severe disease activity), giving an mCPDAI score range of 0 through 12. A higher score indicates more active disease activity. Change from baseline is defined as value at post-baseline visit. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with mCPDAI baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 309 | 306
Score on a scale
  Week 4: number analyzed (Participants) | 305 | 305
  Week 4 | -0.8 (1.57) | -0.7 (1.76)
  Week 8: number analyzed (Participants) | 306 | 303
  Week 8 | -1.3 (1.71) | -0.9 (1.86)
  Week 12 | -1.6 (1.80) | -1.0 (1.87)
  Week 16: number analyzed (Participants) | 303 | 304
  Week 16 | -1.8 (1.97) | -1.2 (2.02)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 4; Test type: Superiority; p = 0.2143, ANCOVA; Adjusted mean difference = -0.2, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.12 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 8; Test type: Superiority; p = 0.0001, ANCOVA; Adjusted mean difference = -0.5, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.13 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -0.7, 95% CI 2-sided [-1.0 to -0.4], Standard Error of Mean 0.13 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Deucravacitinib vs Placebo; Week 16; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -0.6, 95% CI 2-sided [-0.9 to -0.4], Standard Error of Mean 0.14 — [estimate comment as in outcome 2, analysis 1]

34. Secondary Outcome: Number of Participants With Achievement of Psoriatic Arthritis Response Criteria (PsARC)
Description: The Psoriatic Arthritis Response Criteria (PsARC) consists of 4 measurements: tender joint count, swollen joint count, Physician Global Assessment of PsA, and Participant Global Assessment of Disease Activity. In order to be classified as a PsARC responder, participants must achieve improvement in 2 of 4 measures, 1 of which must be joint pain or swelling, without worsening in any measure. Improvement in each of the measures is defined below: 1) Decrease of ≥ 30% in tender joint counts; 2) Decrease of ≥ 30% in swollen joint counts; 3) Decrease of ≥ 20% in Physician Global Assessment of PsA; 4) Decrease of ≥ 20% in Participant's Global Assessment of Disease Activity
Time Frame: Weeks 2, 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 312 | 312
Participants
  Week 2 | 71 | 69
  Week 4 | 128 | 98
  Week 8 | 163 | 126
  Week 12 | 176 | 122
  Week 16 | 187 | 138

35. Secondary Outcome: Number of Participants Meeting Achievement of Improvement of Bath Ankylosing Spondylitis Disease Activity (BASDAI) Score
Description: BASDAI consists of a 0 to 10 scale measuring discomfort, pain, and fatigue in response to 6 questions pertaining to the 5 major symptoms of ankylosing spondylitis: 1) Fatigue (medical); 2) Spinal pain; 3) Joint pain and swelling; 4) Areas of localized tenderness; 5) Morning stiffness duration; 6) Morning stiffness severity. A higher count indicates worse disease. Each individual question response is scaled to a 0-10 score by dividing by 10, and the BASDAI is derived using the following formula: BASDAI = ((Q1 + Q2 + Q3 + Q4) + ((Q5 + Q6) / 2)) / 5
Time Frame: Weeks 2, 4, 8, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with spondylitis in addition to peripheral joint involvement as their presentation of PsA
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 48 | 48
Participants
  Week 2 | 2 | 1
  Week 4 | 6 | 1
  Week 8 | 12 | 5
  Week 12 | 11 | 4
  Week 16 | 17 | 4

36. Secondary Outcome: Change From Baseline in The Work Productivity and Activity Impairment (WPAI) at Week 16
Description: The WPAI is a 6-item questionnaire that includes 2 visual analog scales: 1 for impact of disease on work and 1 for impact of disease on other daily activities. The WPAI also assesses absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity (overall work impairment/absenteeism plus presenteeism), and activity impairment. These sub-scores are transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity. Change from baseline is defined as value at post-baseline visit. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with WPAI baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 306 | 309
Score on a scale
  Absenteeism: number analyzed (Participants) | 183 | 192
  Absenteeism | -0.59 (21.406) | 1.56 (22.108)
  Presenteeism: number analyzed (Participants) | 174 | 183
  Presenteeism | -13.97 (23.380) | -5.96 (22.238)
  Work Productivity: number analyzed (Participants) | 174 | 183
  Work Productivity | -13.71 (24.087) | -5.79 (23.951)
  Activity Impairment | -15.72 (25.226) | -8.16 (24.178)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Absenteeism; Test type: Superiority; p = 0.8316, ANCOVA; Adjusted mean difference = -0.38, 95% CI 2-sided [-3.91 to 3.15], Standard Error of Mean 1.801 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Presenteeism; Test type: Superiority; p = 0.1060, ANCOVA; Adjusted mean difference = -2.95, 95% CI 2-sided [-6.54 to 0.63], Standard Error of Mean 1.827 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Work Productivity; Test type: Superiority; p = 0.1578, ANCOVA; Adjusted mean difference = -2.71, 95% CI 2-sided [-6.47 to 1.05], Standard Error of Mean 1.918 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Deucravacitinib vs Placebo; Activity Impairment; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted mean difference = -7.59, 95% CI 2-sided [-10.96 to -4.22], Standard Error of Mean 1.719 — [estimate comment as in outcome 2, analysis 1]

37. Secondary Outcome: Change From Baseline in the European Quality of Life 5D-5L (EQ-5D-5L) Utility Scores and Its Subcomponents
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. Change from Baseline in 5-level EuroQol 5-dimension (EQ-5D-5L) Utility Scores. Change from baseline is defined as value at post-baseline visit. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Weeks 4, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with EQ-5D-5L baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 307 | 309
Score on a scale
  Week 4 Utility Score: number analyzed (Participants) | 307 | 307
  Week 4 Utility Score | 0.0505 (0.17658) | 0.0655 (0.19080)
  Week 16 Utility Score: number analyzed (Participants) | 306 | 309
  Week 16 Utility Score | 0.0990 (0.21113) | 0.0770 (0.22126)
  Week 4 Mobility: number analyzed (Participants) | 307 | 307
  Week 4 Mobility | -0.2 (0.74) | -0.2 (0.76)
  Week 16 Mobility: number analyzed (Participants) | 306 | 309
  Week 16 Mobility | -0.3 (0.92) | -0.3 (0.87)
  Week 4 Self-Care: number analyzed (Participants) | 307 | 307
  Week 4 Self-Care | -0.1 (0.73) | -0.2 (0.71)
  Week 16 Self-Care: number analyzed (Participants) | 306 | 309
  Week 16 Self-Care | -0.2 (0.83) | -0.2 (0.81)
  Week 4 Usual Activities: number analyzed (Participants) | 307 | 307
  Week 4 Usual Activities | -0.1 (0.76) | -0.2 (0.73)
  Week 16 Usual Activities: number analyzed (Participants) | 306 | 309
  Week 16 Usual Activities | -0.3 (0.84) | -0.3 (0.83)
  Week 4 Pain/Discomfort: number analyzed (Participants) | 307 | 307
  Week 4 Pain/Discomfort | -0.3 (0.75) | -0.3 (0.80)
  Week 16 Pain/Discomfort: number analyzed (Participants) | 306 | 309
  Week 16 Pain/Discomfort | -0.5 (0.89) | -0.4 (0.93)
  Week 4 Anxiety/Depression: number analyzed (Participants) | 307 | 307
  Week 4 Anxiety/Depression | -0.1 (0.76) | -0.1 (0.78)
  Week 16 Anxiety/Depression: number analyzed (Participants) | 306 | 309
  Week 16 Anxiety/Depression | -0.1 (0.77) | 0.0 (0.88)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 4 Utility Score; Test type: Superiority; p = 0.8487, ANCOVA; Adjusted mean difference = -0.0026, 95% CI 2-sided [-0.0291 to 0.0239], Standard Error of Mean 0.01224 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 16 Utility Score; Test type: Superiority; p = 0.0171, ANCOVA; Adjusted mean difference = 0.0365, 95% CI 2-sided [0.0065 to 0.0665], Standard Error of Mean 0.01531 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 4 Mobility; Test type: Superiority; p = 0.9254, ANCOVA; Adjusted mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.06 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Deucravacitinib vs Placebo; Week 16 Mobility; Test type: Superiority; p = 0.0566, ANCOVA; Adjusted mean difference = -0.1, 95% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.06 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Deucravacitinib vs Placebo; Week 4 Self-Care; Test type: Superiority; p = 0.8933, ANCOVA; Ajudted mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.05 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Deucravacitinib vs Placebo; Week 16 Self-Care; Test type: Superiority; p = 0.0738, ANCOVA; Adjusted mean difference = -0.1, 95% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.05 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Deucravacitinib vs Placebo; Week 4 Usual Activities; Test type: Superiority; p = 0.6176, ANCOVA; Adjusted mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.05 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Deucravacitinib vs Placebo; Week 16 Usual Activities; Test type: Superiority; p = 0.1544, ANCOVA; Adjusted mean difference = -0.1, 95% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.06 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Deucravacitinib vs Placebo; Week 4 Pain/Discomfort; Test type: Superiority; p = 0.4707, ANCOVA; Adjusted mean difference = 0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.06 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Deucravacitinib vs Placebo; Week 16 Pain/Discomfort; Test type: Superiority; p = 0.0114, ANCOVA; Adjusted mean difference = -0.2, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.06 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Deucravacitinib vs Placebo; Week 4 Anxiety/Depression; Test type: Superiority; p = 0.6594, ANCOVA; Adjusted mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.05 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: Deucravacitinib vs Placebo; Week 16 Anxiety/Depression; Test type: Superiority; p = 0.7123, ANCOVA; Adjusted mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.06 — [estimate comment as in outcome 2, analysis 1]

38. Secondary Outcome: Change From Baseline in Patient-Reported Outcome Measures Information System (PROMIS)
Description: The Patient-Reported Outcome Measures Information System Sleep Disturbance Short Form 8b assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. The items are evaluated on a 5-point Likert scale ranging from 1 = "not at all" to 5 = "very much" with a 7-day recall period. Higher score means more active disease. Change from baseline is defined as value at post-baseline visit. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Weeks 4, 12, 16
Population: All randomized participants of deucravacitinib and placebo as pre-specified in protocol with PROMIS baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 308 | 309
Score on a scale
  Week 4: number analyzed (Participants) | 307 | 307
  Week 4 | -1.35 (6.958) | -1.41 (6.156)
  Week 12: number analyzed (Participants) | 308 | 306
  Week 12 | -1.76 (7.945) | -1.48 (7.145)
  Week 16: number analyzed (Participants) | 307 | 309
  Week 16 | -2.21 (7.447) | -1.53 (7.134)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Week 4; Test type: Superiority; p = 0.9834, ANCOVA; Adjusted mean difference = -0.01, 95% CI 2-sided [-0.99 to 0.97], Standard Error of Mean 0.498 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Week 12; Test type: Superiority; p = 0.6099, ANCOVA; Adjusted mean difference = -0.29, 95% CI 2-sided [-1.39 to 0.82], Standard Error of Mean 0.565 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Deucravacitinib vs Placebo; Week 16; Test type: Superiority; p = 0.2205, ANCOVA; Adjusted mean difference = -0.66, 95% CI 2-sided [-1.71 to 0.40], Standard Error of Mean 0.538 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed for all participants from date of randomization to their study completion (up to approximately 30 months). SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 30 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Deucravacitinib-Controlled: Deucravacitinib 6 mg daily (Week 0 - Week 16)
- Placebo-Controlled: Placebo daily (Week 0 - Week 16)
- Apremilast-Controlled: Apremilast 30 mg twice daily (Week 0 - Week 16)
- Deucravacitinib-Active Treatment: Deucravacitinib 6 mg daily (Week 16 - Week 52)
- Placebo-Active Treatment: Placebo to Deucravacitinib 6 mg daily (Week 16 - Week 52)
- Apremilast-Active Treatment: Apremilast 30 mg twice daily (Week 16 - Week 52)
- Deucravacitinib-Open Label Extension: Deucravacitinib 6 mg daily (OLE)
- Placebo-Open Label Extension: Placebo to Deucravacitinib 6 mg daily (OLE)
- Apremilast-Open Label Extension: Apremilast 30 mg twice daily (OLE)
Arm/Group | Deucravacitinib-Controlled | Placebo-Controlled | Apremilast-Controlled | Deucravacitinib-Active Treatment | Placebo-Active Treatment | Apremilast-Active Treatment | Deucravacitinib-Open Label Extension | Placebo-Open Label Extension | Apremilast-Open Label Extension
All-Cause Mortality (participants affected / at risk) | 0/312 | 1/312 | 0/105 | 0/292 | 1/292 | 0/90 | 0/245 | 1/254 | 0/70
Serious Adverse Events (participants affected / at risk) | 6/312 | 3/311 | 4/105 | 12/292 | 13/292 | 6/90 | 16/245 | 13/254 | 6/70
Other Adverse Events (participants affected / at risk) | 89/312 | 93/311 | 39/105 | 90/292 | 106/292 | 32/90 | 58/245 | 61/254 | 23/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deucravacitinib-Controlled (N=312) | Placebo-Controlled (N=311) | Apremilast-Controlled (N=105) | Deucravacitinib-Active Treatment (N=292) | Placebo-Active Treatment (N=292) | Apremilast-Active Treatment (N=90) | Deucravacitinib-Open Label Extension (N=245) | Placebo-Open Label Extension (N=254) | Apremilast-Open Label Extension (N=70)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract diabetic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhegmatogenous retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deucravacitinib-Controlled (N=312) | Placebo-Controlled (N=311) | Apremilast-Controlled (N=105) | Deucravacitinib-Active Treatment (N=292) | Placebo-Active Treatment (N=292) | Apremilast-Active Treatment (N=90) | Deucravacitinib-Open Label Extension (N=245) | Placebo-Open Label Extension (N=254) | Apremilast-Open Label Extension (N=70)
Diarrhoea (Gastrointestinal disorders) | 11 | 15 | 11 | 10 | 6 | 11 | 2 | 5 | 3
Nausea (Gastrointestinal disorders) | 7 | 6 | 7 | 5 | 8 | 2 | 3 | 2 | 0
COVID-19 (Infections and infestations) | 22 | 17 | 7 | 19 | 30 | 8 | 13 | 21 | 0
Nasopharyngitis (Infections and infestations) | 14 | 21 | 4 | 27 | 36 | 4 | 14 | 13 | 5
Upper respiratory tract infection (Infections and infestations) | 19 | 13 | 4 | 27 | 28 | 8 | 27 | 16 | 13
Urinary tract infection (Infections and infestations) | 3 | 3 | 2 | 8 | 5 | 5 | 1 | 2 | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 5 | 10 | 2 | 5 | 13 | 5 | 8 | 6 | 2
Headache (Nervous system disorders) | 13 | 11 | 8 | 4 | 4 | 5 | 2 | 3 | 0
Hypertension (Vascular disorders) | 8 | 8 | 7 | 7 | 8 | 0 | 2 | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT04908189/Prot_SAP_000.pdf